CLINICAL TRIAL: NCT02601755
Title: iCanCope With Pain: An Integrated Smartphone and Web Self-management Program for Adolescents and Young Adults With Chronic Pain
Brief Title: iCanCope With Pain: A Smartphone and Web Self-management Program for Adolescents and Young Adults With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Mount Sinai Hospital, Canada (Other); IWK Health Centre (Other); Nova Scotia Health Authority (Other); Stollery Children's Hospital (Other); University of Alberta (Other); Dalhousie University (Other); Centre for Global eHealth Innovation (Other); University of Toronto (Other); University of Saskatchewan (Other); Alberta Children's Hospital (Other); The Ottawa Hospital (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Clinician Scientist, Clinical Nurse Specialist/NP, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000047495
Record Dates: First submitted 2015-11-06; First posted 2015-11-10 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCanCope app and website (Experimental): Intervention: Behavioral: iCanCope app and website
  Interventions: Behavioral: iCanCope app and website
- Attention control group (Active Comparator): Intervention: Behavioral: Attention control group
  Interventions: Behavioral: Attention control group

INTERVENTIONS:
Behavioral: iCanCope app and website — In addition to standard medical care, adolescents and young adults in the experimental group will receive access to the "iCanCope with Pain" smartphone app and website for 8 weeks. The app consists of daily pain symptom tracking (pain intensity, sleep, mood, physical activity, and fatigue), goal setting, in-the moment coping strategies, as well as a social community component. The website provides chronic pain-specific education, self-management strategies, and resources.
  Arms: iCanCope app and website
Behavioral: Attention control group — The control group is designed to control for the potential effects on outcomes of time, attention, smartphone and computer use during the intervention. In addition to standard medical care, adolescents and young adults in the attention control group will receive access to the "iCanCope with Pain" smartphone app (control version, with limited functionality), and a pain resource website without access to self-management strategies.
  Arms: Attention control group

SUMMARY:
Chronic pain in adolescents and young adults (AYA, aged 15-25) is a common problem. Pain that is not treated properly can reduce quality of life. Programs to help AYA learn to live with and manage pain are very important. Our team is developing a smartphone application (app) and website for AYA with chronic pain. The app will help AYA to track pain, sleep, mood, activities, and exercise and help AYA set and achieve goals. The website will give information about pain and how to manage it independently. We will build the program and make sure it is easy to use and understand. We will also test if the program can be put into practice as planned and if AYA using the program feel less pain, have less limitations, and a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic pain of at least 3 months duration according to medical chart
* Able to speak and read English
* Willing and able to complete online measures
* Participants are active patients at pain clinic at one of the respective participating study sites
* Have access to an Internet-connected computer according to self-report.

Exclusion Criteria:

* Moderate to severe cognitive impairments, as assessed by reviewing medical chart and consultation with the patient's healthcare provider
* Major co-morbid psychiatric (e.g. conversion disorder, depression, anxiety disorder) illness that may impact patient's ability to understand and use the iCanCope with Pain intervention via self-report, as determined by their health care provider
* Patient from the department of haemology/oncology
* Participated in the Phase 2B iCanCope usability study
* Requires urgent CBT treatment as per their health care provider
* Individuals who have received more than 4 CBT sessions for pain management in the past 6 months, as per their health-care provider and self-report

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 302 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Participant Accrual and Dropout Rates | 8 weeks
  This will be centrally tracked by the clinical research project coordinator (CRPC).
Intervention fidelity | 8 weeks
  Any issues or difficulties encountered during implementation of the intervention, control strategy, or outcome measures will be tracked throughout the study by the CRPC.
Acceptability and Satisfaction | 8 weeks
  Participants in the intervention arm will complete the Acceptability e-scale (AES) post-intervention. In addition, a subset of participants from the intervention group will be offered to participate in a qualitative feedback interview to further explore acceptability and satisfaction of the intervention.
Engagement with Intervention | 8 weeks
  Google Analytics will track patterns of app and website usage.
Adherence | 8 weeks
  Adherence will be determined using Google Analytics.

SECONDARY OUTCOMES:
Pain intensity and interference | 8 weeks
  Measured using the short form Brief Pain Inventory (BPI), a 15-item tool that measures pain intensity and impact on functioning.
Self-efficacy | 8 weeks
  Measured with the Pain Self-Efficacy Questionnaire (PSEQ), a 10-item scale that requires patients to take their pain into account when rating their self-efficacy beliefs.
Emotional Functioning | 8 weeks
  Measured using the Hospital Anxiety and Depression Scale (HADS), a 14-item measure for the assessment of anxiety and depressive symptoms.
Sleep Functioning | 8 weeks
  Measured with the Insomnia Severity Index (ISI), a 7-item self-report questionnaire for assessing the nature, severity, and impact of insomnia.
Social Functioning | 8 weeks
  Measured with the Perceived Social Support from Friends (PSS-Fr) Scale, a 20-item scale that assesses the extent to which an individual perceives that their friends fulfill their needs for support.
Health-Related Quality of Life | 8 weeks
  Measured using the SF-36 Health Survey, a 36-item self-report scale with 8 subscales (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health).
Patients' Global Impression of Change | 8 weeks
  Measured using the PGIC scale, a single item rating by participants of their perceived change during the trial.
Pain-Related Knowledge | 8 weeks
  Measured using a modified version of the Medical Issues, Exercise, Pain and Social Support (MEPS) questionnaire, a 27-item measure.
Health Care Utilization | 8 weeks
  Measured using the Chronic Pain Healthcare Utilization Form. (modified from the Ambulatory and Home Care Record)
Adverse effects | 8 weeks
  Will be tracked using the adverse event form.

CONTACTS AND LOCATIONS:
Locations (10):
- Canada (10):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - Nova Scotia Health Authority/Dalhousie University, Halifax, Nova Scotia
  - IWK Health Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Lalloo C, Hundert A, Harris L, Pham Q, Campbell F, Chorney J, Dick B, Simmonds M, Cafazzo J, Stinson J. Capturing Daily Disease Experiences of Adolescents With Chronic Pain: mHealth-Mediated Symptom Tracking. JMIR Mhealth Uhealth. 2019 Jan 17;7(1):e11838. doi: 10.2196/11838. PMID 30664472